CLINICAL TRIAL: NCT02439151
Title: New Lung Ventilation Strategies Guided by Transpulmonary Pressure in VV-ECMO for Severe ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rui Wang (Other)
Responsible Party: Sponsor-Investigator, Rui Wang, Principal Investigator, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-KE-143
Record Dates: First submitted 2015-05-01; First posted 2015-05-08 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Extracorporeal Membrane Oxygenation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- New Strategy (Experimental): New Strategy: use transpulmonary pressure guide new lung ventilation strategy in ECMO for severe ARDS patients
  Interventions: Device: New lung ventilation strategy
- Conventional Strategy (Other): Conventional Strategy: use conventional ventilation strategy (ELSO guide ventilation strategy) in ECMO for severe ARDS patients
  Interventions: Device: Conventional ventilation strategy

INTERVENTIONS:
Device: New lung ventilation strategy — New ventilation strateg: pressure assist control mode; inspiratory pressure was lowered to keep Ppeak less than 25cmH2O; set the PEEP at such a level that expiratory transpulmonary pressure stays between 0 and 5 cmH2O; respiratory rate of 10 breaths per minute; FiO2 less than 0.5.
  Arms: New Strategy
Device: Conventional ventilation strategy — Conventional ventilation strategy: pressure assist control mode; keep the Ppeak between 20 and 25 cmH2O; set PEEP between 10 and 15 cmH2O; respiratory rate of 10 breaths per minute; FiO2 less than 0.5.
  Arms: Conventional Strategy

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) has been widely used in patients with severe acute respiratory distress syndrome (ARDS). But how to choose mechanical ventilation strategy is still not clear for severe ARDS patients supported by ECMO. Our previous work found that, compared to the traditional "lung rest" strategy, transpulmonary pressure guide new lung ventilation strategy can better maintain lung volume reduction lung collapse, atelectasis occurs. The severe ARDS patients receiving ECMO therapy were randomized divided into a new ventilation strategy group and the conventional ventilation strategy group. The new ventilation strategy is transpulmonary pressure guide ventilator setting method, and the conventional ventilation strategy is Extracorporeal Life Support Organization (ELSO) guide ventilation method. Compare the difference between the two groups of patients in lung injury, and explore the lung protection mechanism of new lung ventilation strategies guided by transpulmonary pressure. Our research group considered that transpulmonary pressure guide new lung ventilation strategy can provide more effective lung protection. And it will be further used in clinical work.

ELIGIBILITY:
Inclusion Criteria:

* ARDS cause reversible;
* Pure oxygen is given, but PaO2/FiO2<80;
* P(A-a)O2>600mmHg;
* Murray score≥3.0;
* pH<7.2;

Exclusion Criteria:

* peak inspiratory pressure>30cmH2O;
* high FiO2>0.8;
* ventilation>7 days;
* contraindication to heparinization;
* non-reversible central nervous system injury
* chronic disease with a short life expectancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Proportion weaned from VV-ECMO | After patients randomized grouping 60 days
  Respiratory failure was alleviated and then ECMO withdrawal could be considered

SECONDARY OUTCOMES:
60-day mortality | After patients randomized grouping 60 days
  Mortality after patients randomized grouping 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Bing Sun, master, Principal Investigator — Beijing Chao-Yang Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China